CLINICAL TRIAL: NCT00574977
Title: A Phase I Dose-escalation Trial of vvDD-CDSR (Double-deleted Vaccinia Virus Plus CD/ SMR) Administered by Intratumoral Injection or Intravenous Injection
Brief Title: Safety Study of Modified Vaccinia Virus to Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Bartlett (Other)
Responsible Party: Sponsor-Investigator, David Bartlett, Chief, Division of Surgical Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-041
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Melanoma; Breast Cancer; Head and Neck Squamous Cell Cancer; Liver Cancer; Colorectal Cancer; Pancreatic Adenocarcinoma
Keywords: vaccinia; virus; tumor; melanoma; breast cancer; squamous cell cancer; colorectal; liver; pancreatic; adenocarcinoma
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Liver Neoplasms; Colorectal Neoplasms; Vaccinia; Virus Diseases; Neoplasms; Neoplasms, Squamous Cell; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Subjects who have been vaccinated with vaccinia virus (small pox)and will receive vvDD-CDSR by intratumoral injection
  Interventions: Biological: Vaccinia virus (vvDD-CDSR)
- B (Experimental): Subjects will include those who have not been vaccinated with vaccinia virus (small pox)and will receive vvDD-CDSR by intratumoral injection.
  Interventions: Biological: Vaccinia virus (vvDD-CDSR)
- C (Experimental): Subjects will be those who have been vaccinated with vaccinia virus (small pox)and will be receiving the vvCD-CDSR via intravenous infusion
  Interventions: Biological: Vaccinia virus (vvDD-CDSR)

INTERVENTIONS:
Biological: Vaccinia virus (vvDD-CDSR) — Eligible subjects will receive 1 treatment of vvDD-CDSR. A dose can be divided between 1-3 lesions. The sum total of the maximal diameters of the lesion(s) to be injected must be < 10cm.
  Cohort 1: 3 x 10e7 p.f.u. Cohort 2: 1 x 10e8 p.f.u. Cohort 3: 3 x 10e8 p.f.u. Cohort 4: 1 x 10e9 p.f.u. Cohort 5: 3 x 10e9 p.f.u.
  Arms: A
Biological: Vaccinia virus (vvDD-CDSR) — Eligible subjects will receive 1 treatment of vvDD-CDSR. A dose can be divided between 1-3 lesions. The sum total of the maximal diameters of the lesion(s) to be injected must be < 10cm.
  Cohort 1: 3 x 10e7 p.f.u. Cohort 2: 1 x 10e8 p.f.u. Cohort 3: 3 x 10e8 p.f.u. Cohort 4: 1 x 10e9 p.f.u. Cohort 5: 3 x 10e9 p.f.u.
  Arms: B
Biological: Vaccinia virus (vvDD-CDSR) — Eligible subjects will receive 1 infusion of vvDD-CDSR.
  Cohort 1: 3 x 10e8 p.f.u; Cohort 2: 1 x 10e9 p.f.u.; Cohort 3: 3 x 10e9 p.f.u.
  Arms: C

SUMMARY:
The purpose of this study is to determine the safety and maximum tolerated dose from injecting this vaccinia virus into tumors or infusion.

DETAILED DESCRIPTION:
This is a Phase I, open-label, single dose, dose-escalation trial in subjects with melanoma, breast cancer, or head and neck squamous cell cancer, liver, colorectal or pancreatic adenocarinoma. The intratumoral subjects will be stratified into 2 groups. Group A includes those who have been vaccinated with vaccinia virus. A history of vaccination and a scar at vaccination site is required. Group B subjects will include those who have not been vaccinated. It is expected that the toxicity profile will be quite different between those who have been vaccinated previously with vaccinia virus and therefore subjects will be stratified separately in this Phase I trial. All subjects who have refractory tumors will receive treatment at one of five dose levels in a single dose sequential dose-escalating design. Eligible subjects will receive 1 treatment of vvDD-CDSR. A dose can be divided between 1-3 lesions. The sum total of the maximal diameters of the lesion(s) to be injected must be < 10cm.

Once the MTD and/or MFD has been defined in the vaccinated I.T. arm described above, additional subject may be enrolled at one dose level lower than the MTD/MFD and the I.V. infusion phase may begin. Patients enrolled in the IV infusion arm will receive a single administration of vvDD-CDSR at one of three dose levels in a sequential dose-escalating design.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Histologically-confirmed cancer that has progressed despite standard therapy. They must have one of the following tumor-types: melanoma, breast cancer, or head and neck squamous cell cancer, liver, colorectal or pancreatic
* Cancer is not surgically curable
* Karnofsky Performance Status (KPS) of > 70 (See Appendix B)
* Anticipated survival of at least 16 weeks
* If sexually-active, willingness to use condoms for 3 months following study treatment with vvDD-CDSR
* The ability to understand and willingness to sign a written informed consent
* Able to comply with study procedures and follow-up examinations
* Adequate bone marrow function: WBC > 3,500 and <50,000 cells/mm3, ANC > 1,500 cells/mm3, hemoglobin > 10 g/dL, and platelet count > 150,000 cells/mm3
* Adequate renal function: serum creatinine level ≤ 1.2 x ULN

Exclusion Criteria:

* Pregnant or nursing an infant
* Active viral infection (including HIV, Hepatitis B and C)
* Systemic corticosteroid or other immunosuppressive medication use within 4 weeks of the treatment
* Clinically significant active infection or uncontrolled medical condition (e.g., pulmonary, neurological, cardiovascular, gastrointestinal, genitourinary) considered high risk for investigational new drug treatment
* Significant immunodeficiency (e.g. due to underlying illness and/ or medication) in subject or household contacts
* History of eczema requiring systemic therapy
* Unstable cardiac disease which includes but is not limited to: Any of the following within 6 months prior to study entry: MI, unstable angina, congestive heart failure, myocarditis, arrhythmias diagnosed and requiring medication, or any clinically-significant change in cardiac status
* Target tumor(s) adherent to a major vascular structure (e.g. carotid artery)
* Subjects who have received radiation, chemotherapy or other potentially immunosuppressive therapy in 4 weeks prior to study screening
* Clinically significant and/or rapidly accumulating ascites, peri-cardial and/or pleural effusions
* Experienced a severe systemic reaction or side-effect as a result of a previous smallpox vaccination
* Subjects with household contacts who are pregnant or nursing an infant, children < 5 years old, have history of eczema that at some stage has required systemic therapy, or have a significant immunodeficiency due to underlying illness (e.g. HIV) and/or medication (e.g. systemic corticosteroids) will be excluded unless alternate living arrangements can be made during the subject's active dosing period and for three weeks following the last dose of study medication
* Inability or unwillingness to give informed consent.
* CD4 T cell count < 350 per µL blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-05; Primary Completion 2013-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximally tolerated dose (MTD) and/or maximum-feasible dose (MFD) and Safety of vvDD-CDSR administered by intratumoral (I.T.) injection and intravenous (I.V.) infusion. | 28 days

SECONDARY OUTCOMES:
Replication/pharmacokinetics of vvDD-CDSR | 28 days
Immune response to vvDD-CDSR and to the tumor following administration | 28 days
Antitumoral efficacy of vvDD-CDSR | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert J. Zeh, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States